CLINICAL TRIAL: NCT02682381
Title: A 24-Week Double-blind, Safety, Efficacy, and Pharmacodynamic Study Investigating Two Doses of Teduglutide in Pediatric Subjects Through 17 Years of Age With Short Bowel Syndrome Who Are Dependent on Parenteral Support
Brief Title: Short Bowel Syndrome Research Study for Children Up To 17 Years of Age on Parenteral Nutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TED-C14-006
Record Dates: First submitted 2016-01-27; First posted 2016-02-15 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: Teduglutide; pediatric; GLP-2; parenteral support; Short Bowel Syndrome; short gut syndrome; short gut; SBS; parenteral nutrition
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — teduglutide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.025 mg/kg/day Teduglutide (Experimental): 0.025 milligrams per kilogram per day (mg/kg/day) of teduglutide for 24 weeks.
  Interventions: Drug: Teduglutide 0.025 mg/kg
- 0.05 mg/kg/day Teduglutide (Experimental): 0.05 mg/kg/day of teduglutide for 24 weeks.
  Interventions: Drug: Teduglutide 0.05mg/kg
- Standard of care (Active Comparator): Observational cohort for the 24-week treatment period and 4 week follow-up. The subjects in the standard of care group will follow the same visit schedule as the randomized subjects.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Teduglutide 0.05mg/kg — 0.05 mg/kg
  Arms: 0.05 mg/kg/day Teduglutide
Drug: Teduglutide 0.025 mg/kg — 0.025 mg/kg
  Arms: 0.025 mg/kg/day Teduglutide
Other: Standard of Care — Observational cohort for the 24-week treatment period and 4 week follow-up.
  Arms: Standard of care

SUMMARY:
Teduglutide is approved for treatment of adults with short bowel syndrome (SBS). The purpose of this study is to evaluate the safety and efficacy of teduglutide in children up to the age of 17 with SBS who are dependent on parenteral support. Subjects may choose whether to receive the study drug or to participate in a standard-of-care arm. All participants who complete the study may be eligible to receive the study drug in a long-term extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent by a parent or guardian or emancipated minor prior to any study-related procedures
2. When applicable, an informed assent by the subject (as deemed appropriate by the Ethics Committee/Institutional Review Board) prior to any study-related procedures
3. Current history of SBS as a result of major intestinal resection, (eg, due to necrotizing enterocolitis, midgut volvulus, intestinal atresia, or gastroschisis)
4. Short bowel syndrome that requires PN/IV support that provides at least 30% of caloric and/or fluid/electrolyte needs prior to screening
5. Stable PN/IV support, defined as inability to significantly reduce PN/IV support, usually associated with minimal or no advance in enteral feeds (ie, 10% or less change in PN or advance in feeds) for at least 3 months prior to and during screening, as assessed by the investigator.
6. Sexually active female subjects of child-bearing potential (in the teduglutide treatment arm only) must use medically acceptable methods of birth control during and 4 weeks after the treatment period

Exclusion Criteria:

1. Subjects who are not expected to be able to advance oral or tube feeding regimens
2. Serial transverse enteroplasty or any other bowel lengthening procedure performed within 3 months of screening
3. Known clinically significant untreated intestinal obstruction contributing to feeding intolerance and inability to reduce parenteral support
4. Unstable absorption due to cystic fibrosis or known DNA abnormalities
5. Severe, known dysmotility syndrome, such as pseudo-obstruction or persistent, severe, active gastroschisis-related dysmotility, that is the primary contributing factor to feeding intolerance and inability to reduce parenteral support, prior to screening. Dysmotility is defined as severe if it is expected to limit the advancement of enteral feeding.
6. Evidence of clinically significant obstruction on upper GI series done within 6 months prior to screening.
7. Major GI surgical intervention including significant intestinal resection within 3 months prior to the screening visit (insertion of feeding tube, anastomotic ulcer repair, minor intestinal resections ≤ 10 cm, or endoscopic procedure is allowed).
8. Unstable cardiac disease, congenital heart disease or cyanotic disease, with the exception of subjects who had undergone ventricular or atrial septal defect repair, and patent ductus arteriosus (PDA) ligation.
9. History of cancer or clinically significant lymphoproliferative disease, not including resected cutaneous basal or squamous cell carcinoma, or in situ non aggressive and surgically resected cancer.
10. Pregnant or lactating female subjects (in the teduglutide treatment arm only).
11. Participation in a clinical study using an experimental drug (other than glutamine or Omegaven) within 3 months or 5.5 half-lives of the experimental drug, whichever is longer, prior to screening, and for the duration of the study.
12. Previous use of teduglutide or native/synthetic glucagon-like peptide-2 (GLP-2)
13. Previous use of glucagon-like peptide-1 analog or human growth hormone within 3 months prior to screening
14. Previous use of octreotide, or dipeptidyl peptidase-4 (DPP-4) inhibitors within 3 months prior to screening
15. Subjects with active Crohn's disease who had been treated with biological therapy (eg, antitumor necrosis factor [anti-TNF]) within the 6 months prior to the screening visit
16. Subjects with inflammatory bowel disease (IBD) who require chronic systemic immunosuppressant therapy that had been introduced or changed during the 3 months prior to screening
17. More than 3 SBS-related or PN-related hospital admissions (eg, documented infection-related catheter sepsis, clots, bowel obstruction, severe water-electrolyte disturbances) within 3 months prior to the screening visit
18. Any major unscheduled hospital admission which affects parenteral support requirements within 1 month prior to or during screening, excluding uncomplicated treatment of bacteremia, central line replacement/repair, or issues of similar magnitude in an otherwise stable subject
19. Body weight < 10 kg at the screening and baseline visits
20. Signs of active severe or unstable, clinically significant hepatic impairment during the screening period, as indicated by any of the following laboratory test results :

    1. Total bilirubin (TBL) ≥ 2 x upper limit of normal (ULN)
    2. Aspartate aminotransferase (AST) ≥ 7x ULN
    3. Alanine aminotransferase (ALT) ≥ 7x ULN

       For subjects with Gilbert's disease:
    4. Indirect (unconjugated) bilirubin ≥ 2x ULN
21. Signs of known continuous active or unstable, clinically significant renal dysfunction shown by results of an estimated glomerular filtration rate (eGFR) below 50 mL/min/1.73 m2.
22. Parent(s) and/or subjects who are not capable of understanding or not willing to adhere to the study visit schedule and other protocol requirements
23. Unstable, clinically significant active, untreated pancreatic or biliary disease
24. Any condition, disease, illness, or circumstance that in the investigator's opinion puts the subject at any undue risk, prevents completion of the study, or interferes with analysis of the study results.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- United States (18):
  - Children's Hospital Los Angeles - RHU, Los Angeles, California
  - UCLA Dept. of Medicine, Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Georgetown Children's Research Network, Washington D.C., District of Columbia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - The Nebraska Medical Center, Omaha, Nebraska
  - Children's Hospital GI Nutrition, New York, New York
  - Montefiore Medical Center Child Spc, The Bronx, New York
  - Duke Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Pediatric Specialists, Cleveland, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Canada (3):
  - Walter C. Mackenzie Health Science Center, Edmonton, Alberta
  - British Columbia Children's & Women's Hospital Center, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
- Helsingin yliopistollinen keskussairaala, Helsinki, Finland
- Universitaetsklinikum Tuebingen, Tübingen, Baden Wuertternberg, Germany
- Ospedale Pediatrico Bambino Gesu, Roma, Italy
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London, Greater London
  - Birmingham Children's Hospital, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Fifi A, Raphael BP, Terreri B, Uddin S, Kaufman SS. Effects of Teduglutide on Diarrhea in Pediatric Patients with Short Bowel Syndrome-Associated Intestinal Failure. J Pediatr Gastroenterol Nutr. 2023 Nov 1;77(5):666-671. doi: 10.1097/MPG.0000000000003922. Epub 2023 Aug 22. PMID 37889619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 27 study centers in the United States, Belgium, Canada, the United Kingdom, Finland, Germany and Italy between 03 June 2016 (first participant first visit) and 18 August 2017 (last participant last visit).
Pre-assignment Details: Overall, 59 participants were enrolled; 50 in the teduglutide treatment arm (24 participants in the 0.025 milligram per kilogram per day (mg/kg/day) dose group and 26 participants in the 0.05 mg/kg/day dose group)and 9 in the standard of care arm.
Groups:
- 0.025 mg/kg/Day Teduglutide: Participants received 0.025 milligram per kilogram per day (mg/kg/day) of teduglutide subcutaneously for 24 weeks along with standard medical therapy.
- 0.05 mg/kg/Day Teduglutide: Participants received 0.05 mg/kg/day of teduglutide subcutaneously for 24 weeks along with standard medical therapy.
- Standard of Care: Participants received standard medical therapy.
Period: Overall Study
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Started | 24 | 26 | 9
Completed | 24 | 26 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all enrolled participants.
Groups:
- 0.025 mg/kg/Day Teduglutide: Participants received 0.025 mg/kg/day of teduglutide subcutaneously for 24 weeks along with standard medical therapy.
- Total: Total of all reporting groups
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care | Total
Number analyzed (Participants) | 24 | 26 | 9 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (3.61) | 6.2 (3.67) | 5.7 (4.72) | 6.3 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 3 | 18
  Male | 16 | 19 | 6 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 4 | 14
  Not Hispanic or Latino | 16 | 20 | 2 | 38
  Unknown or Not Reported | 3 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Customized race population was reported here.
  Participants
    Race Customized: White | 16 | 21 | 2 | 39
    Race Customized: Black or African American | 3 | 3 | 1 | 7
    Race Customized: Asian | 1 | 1 | 1 | 3
    Race Customized: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Race Customized: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Race Customized: Other | 1 | 0 | 2 | 3
    Race Customized: Not allowed based on local regulations | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved at Least a 20 Percent (%) Reduction in Weight-Normalized Average Daily Parenteral Nutrition Intravenous (PN/IV) Volume at Week 24
Description: Reduction in weight-normalized PN/IV volume was performed using both participant diary and investigator prescribed data. Number of participants who achieved at least a 20% reduction in weight-normalized PN/IV volume between the baseline and week 24/EOT visit were reported.
Time Frame: Baseline through Week 24
Population: ITT population included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Participants
  Participant Diary | 13 | 18 | 1
  Investigator Prescribed | 13 | 18 | 2

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that started or worsened on or after the date of first dose for treatment groups and those that started or worsened on or after the baseline visit for standard of care group.
Time Frame: From start of study treatment up to 28 weeks
Population: Safety analysis population included all participants who received at least 1 dose of teduglutide and had undergone at least 1 post-baseline safety assessment in teduglutide treatment group or participants who had undergone at least 1 post-baseline safety assessment in standard of care treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Participants | 24 | 25 | 9

3. Secondary Outcome: Number of Participants Who Were Completely Weaned Off Parenteral Nutrition Intravenous (PN/IV) Support at Week 24
Description: A participant was considered to have achieved independence from PN/IV support (completely weaned off PN/IV) if the investigator prescribed no PN/IV at EOT and there was no use of PN/IV recorded in the participant diary during the week prior to EOT.
Time Frame: Week 24
Population: ITT population included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Participants | 2 | 3 | 0

4. Secondary Outcome: Change From Baseline in Parenteral Nutrition Intravenous (PN/IV) Volume at Week 24
Description: Change in PN/IV volume was reported based on the participant diary and the investigator prescribed data.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Milliliters per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Milliliters per kilogram per day
  Participant Diary: number analyzed (Participants) | 20 | 25 | 9
  Participant Diary | -16.16 (10.52) | -23.30 (17.50) | -6.03 (4.55)
  Investigator Prescribed | -11.28 (15.51) | -22.13 (17.92) | -5.84 (9.80)

5. Secondary Outcome: Change From Baseline in Parenteral Nutrition Intravenous (PN/IV) Caloric Intake at Week 24
Description: Change in PN/IV caloric intake was reported based on the participant diary and the investigator prescribed data.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Kilocalories per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Kilocalories per kilogram per day
  Participant Diary: number analyzed (Participants) | 20 | 25 | 9
  Participant Diary | -14.92 (8.29) | -18.99 (14.28) | -0.46 (4.95)
  Investigator Prescribed: number analyzed (Participants) | 24 | 25 | 9
  Investigator Prescribed | -11.76 (10.46) | -18.51 (13.22) | -0.27 (2.73)

6. Secondary Outcome: Change From Baseline in Plasma Citrulline Levels at Week 24
Description: Plasma citrulline level was reported.
Time Frame: Baseline, Week 24
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 21 | 24 | 8
Micromoles per liter | 7.7 (8.50) | 12.0 (12.00) | 0.1 (7.79)

7. Secondary Outcome: Change From Baseline in Enteral Nutrition Volume at Week 24
Description: Enteral nutrition was defined as specialized formula taken orally or by tube feeding, and excluded table foods and other fluids. Change in enteral nutrition volume was reported.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Milliliter per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Milliliter per kilogram per day
  Participant Diary: number analyzed (Participants) | 18 | 25 | 9
  Participant Diary | 7.69 (13.46) | 10.96 (16.59) | 0.74 (5.91)
  Investigator Prescribed: number analyzed (Participants) | 18 | 21 | 5
  Investigator Prescribed | 7.67 (17.77) | 8.17 (17.87) | 0.33 (0.90)

8. Secondary Outcome: Change From Baseline in Enteral Nutrition Caloric Intake at Week 24
Description: Enteral nutrition was defined as specialized formula taken orally or by tube feeding, and excluded table foods and other fluids. Change in enteral nutrition caloric intake was reported.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Kilocalorie per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Kilocalorie per kilogram per day
  Participant Diary: number analyzed (Participants) | 18 | 25 | 9
  Participant Diary | 8.43 (14.39) | 12.98 (18.93) | 4.22 (13.75)
  Investigator Prescribed: number analyzed (Participants) | 18 | 21 | 5
  Investigator Prescribed | 7.29 (15.88) | 11.47 (21.13) | 6.66 (14.77)

9. Secondary Outcome: Change From Week 24 in Parenteral Nutrition Intravenous (PN/IV) Volume at Week 28
Description: Change in PN/IV volume was reported.
Time Frame: Week 24, Week 28
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Milliliter per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Milliliter per kilogram per day
  Participant Diary: number analyzed (Participants) | 24 | 26 | 8
  Participant Diary | 2.63 (7.80) | 1.52 (12.68) | -2.99 (4.94)
  Investigator Prescribed | 2.13 (6.95) | -0.35 (5.96) | -0.91 (2.18)

10. Secondary Outcome: Change From Week 24 in Parenteral Nutrition Intravenous (PN/IV) Caloric Intake at Week 28
Description: Change in PN/IV caloric intake was reported.
Time Frame: Week 24, Week 28
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Kilocalorie per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Kilocalorie per kilogram per day
  Participant Diary: number analyzed (Participants) | 24 | 26 | 8
  Participant Diary | 0.88 (2.94) | -0.91 (7.14) | -4.21 (10.30)
  Investigator Prescribed | 0.55 (3.42) | 0.08 (6.13) | -4.34 (11.22)

11. Secondary Outcome: Change From Week 24 in Plasma Citrulline Levels at Week 28
Description: Change in plasma citrulline level was reported.
Time Frame: Week 24, Week 28
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 25 | 9
Micromoles per liter | -6.0 (9.26) | -9.5 (10.33) | 1.8 (6.48)

12. Secondary Outcome: Change From Week 24 in Enteral Nutrition Volume at Week 28
Description: as for outcome 7
Time Frame: Week 24, Week 28
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Milliliter per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Milliliter per kilogram per day
  Participant Diary: number analyzed (Participants) | 23 | 26 | 8
  Participant Diary | -0.68 (3.86) | 1.38 (8.41) | -0.75 (6.78)
  Investigator Prescribed: number analyzed (Participants) | 18 | 22 | 5
  Investigator Prescribed | 1.67 (5.73) | 0.68 (6.65) | 0.39 (0.57)

13. Secondary Outcome: Change From Week 24 in Enteral Nutrition Caloric Intake at Week 28
Description: as for outcome 8
Time Frame: Week 24, Week 28
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Kilocalorie per kilogram per day
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Kilocalorie per kilogram per day
  Participant Diary: number analyzed (Participants) | 23 | 26 | 8
  Participant Diary | -1.07 (4.36) | -0.14 (7.73) | -0.42 (6.13)
  Investigator Prescribed: number analyzed (Participants) | 18 | 22 | 5
  Investigator Prescribed | 1.28 (4.30) | -0.11 (3.77) | 0.45 (0.64)

14. Secondary Outcome: Change From Baseline in Body Weight Z-score at Week 28
Description: Body weight z-score is a measure of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline, Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Z-score | -0.12 (0.41) | -0.18 (0.59) | -0.05 (0.37)

15. Secondary Outcome: Change From Baseline in Body Height Z-score at Week 28
Description: Body height z-score is a measure of relative height adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline, Week 28
Population: Safety analysis population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 25 | 9
Z-score | 0 (0.29) | 0.05 (0.45) | 0.16 (0.66)

16. Secondary Outcome: Change From Baseline in Head Circumference Z-score at Week 28
Description: Head circumference z-score is a measure of relative head circumference adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. Head circumference was collected only for participants of less than or equal to (<=) 36 months of age at the time of measurement.
Time Frame: Baseline, Week 28
Population: Safety analysis population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 0 | 0 | 1
Z-score |  |  | -0.014 (NA) — "NA" signifies that the standard deviation was not calculated due to less number of participants.

17. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Z-score at Week 28
Description: BMI z-score is a measure of relative BMI adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline, Week 28
Population: Safety analysis population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 25 | 9
Z-score | -0.13 (0.57) | -0.22 (0.70) | -0.25 (1.42)

18. Secondary Outcome: Change From Baseline in Participants' Stool Consistency at Week 28
Description: Stool consistency was assessed by typical stool form based on Bristol Stool Form Scale: 1 - Separate hard lumps, hard to pass, 2 - Sausage-shaped, but lumpy, 3 - Like a sausage but with cracks on the surface, 4 - Like a sausage or snake, smooth and soft, 5 - Soft blobs with clear-cut edges, 6 - Fluffy pieces with ragged edges, a mushy stool, 7 - Watery, no solid pieces, entirely liquid.
Time Frame: Baseline, Week 28
Population: Safety analysis population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 8 | 16 | 2
Score on a scale | -1.3 (1.77) | -1.4 (1.38) | -3.3 (0.35)

19. Secondary Outcome: Change From Baseline in Hours Per Day of Parenteral Nutrition Intravenous (PN/IV) Support at Week 24
Description: The mean duration of the PN/IV infusions in hours, on the days when PN/IV was administered was reported.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Hours per day (hour/day)
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Hours per day (hour/day)
  Participant Diary: number analyzed (Participants) | 22 | 26 | 9
  Participant Diary | -2.47 (2.73) | -3.03 (3.84) | -0.21 (0.69)
  Investigator Prescribed | -1.48 (3.59) | -1.79 (3.52) | 0.11 (0.33)

20. Secondary Outcome: Change From Baseline in Days Per Week of Parenteral Nutrition Intravenous (PN/IV) Support at Week 24
Description: The number of days per week of PN/IV infusions were reported.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Days per week (Days/week)
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
Number analyzed (Participants) | 24 | 26 | 9
Days per week (Days/week)
  Participant Diary: number analyzed (Participants) | 22 | 26 | 9
  Participant Diary | -0.88 (1.78) | -1.34 (2.24) | 0 (0)
  Investigator Prescribed | -0.79 (1.62) | -1.42 (2.32) | 0 (0)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 28 weeks
Arm/Group | 0.025 mg/kg/Day Teduglutide | 0.05 mg/kg/Day Teduglutide | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26 | 0/9
Serious Adverse Events (participants affected / at risk) | 15/24 | 20/26 | 4/9
Other Adverse Events (participants affected / at risk) | 24/24 | 23/26 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.025 mg/kg/Day Teduglutide (N=24) | 0.05 mg/kg/Day Teduglutide (N=26) | Standard of Care (N=9)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 7 (8) | 1 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (2) | 3 (3) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 2 (3) | 2 (2) | 0 (0) — TEAEs coded to Product issues were related to central line complications, and not due to complications of the investigational product and ancillary supplies.
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) — TEAEs coded to Product issues were related to central line complications, and not due to complications of the investigational product and ancillary supplies.
Device issue (Product Issues) | 0 (0) | 1 (1) | 0 (0) — TEAEs coded to Product issues were related to central line complications, and not due to complications of the investigational product and ancillary supplies.
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) — TEAEs coded to Product issues were related to central line complications, and not due to complications of the investigational product and ancillary supplies.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.025 mg/kg/Day Teduglutide (N=24) | 0.05 mg/kg/Day Teduglutide (N=26) | Standard of Care (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 6 (7) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (8) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 10 (23) | 8 (17) | 5 (7)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 2 (2)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 3 (4) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 6 (9) | 3 (4)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 2 (6) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (9) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 1 (1) | 5 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 6 (8) | 4 (5)
Urinary tract infection (Infections and infestations) | 2 (4) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 3 (4) | 1 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 4 (5) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 2 (2) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Drug-Induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (9) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (4) | 5 (7) | 1 (3)
Device breakage (Product Issues) | 2 (2) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (11) | 3 (4)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (20) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonmentor termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Protocol (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT02682381/Prot_000.pdf
  • Study Protocol: Amendment1 (2015-06-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT02682381/Prot_001.pdf
  • Study Protocol: Amendment3 (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02682381/Prot_002.pdf
  • Study Protocol: Amendment4 (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02682381/Prot_003.pdf
  • Study Protocol: Amendment2 (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT02682381/Prot_005.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT02682381/SAP_004.pdf